CLINICAL TRIAL: NCT05796336
Title: Effectiveness of Two Methods of Lip Taping as a Presurgical Orthopedic in Infants With Bilateral Cleft Lip and Palate: A Randomized Clinical Trial
Brief Title: Two Methods of Lip Taping as a Presurgical Orthopedic Appliance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Mushriq F. Abid, Professor, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 765423
Record Dates: First submitted 2023-03-18; First posted 2023-04-03 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive lip taping (Experimental): Will receive passive baby feeding plate and conventional steri strip
  Interventions: Device: Lip taping
- Custom-made tape (Experimental): will receive passive baby feeding plate and custom-made tape (Steri Srip and orthodontic elastics)
  Interventions: Device: Lip taping

INTERVENTIONS:
Device: Lip taping — Steri strip tape and passive baby feeding plate Two methods of lip taping will be used with passive baby feeding plate. Impressions will be taken before starting the treatment (T1) and at the end of treatment (T2) three months later. The effectiveness of the two appliances will be assessed and measured on digital models of the maxillary arch before and after the treatment.

SUMMARY:
A randomized clinical trial to compare the effectiveness of two methods of lip taping as a presurgical orthopedic appliances on maxillary arch dimensions in infants with bilateral cleft lip and palate.

DETAILED DESCRIPTION:
It is a multicenter randomized clinical trial with two parallel arms. The patients will be randomly divided into two groups, group one: a passive orthopedic appliance will be used with conventional steri strip, and group two will receive a passive orthopedic appliance with a custom-made tape consist of steri strip and orthodontic elastic. Impressions will be taken before starting the treatment (T1) and at the end of treatment (T2) three months later. The effectiveness of the two methods of taping will be assessed and measured on digital models of the maxillary arch before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Non-Syndromic infants with complete bilateral cleft lip and palate.
2. Both sexes.
3. Age range from 1-30 day

Exclusion Criteria:

1. Infants with systemic syndromes.
2. infants with unilateral cleft
3. infants whom parents refuse to consent.

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of maxillary arch dimension change | T1 before starting any treatment and T2 After treatment before surgical repair (average 3 months)]
  To evaluate the effect of the lip taping as a presurgical orthopedic on the maxillary arch dimensions for infants with bilateral cleft using two different types of medical taping.

SECONDARY OUTCOMES:
Assessment of Linear measurement change | T1 before starting any treatment and T2 After treatment before surgical repair (average 3 months)]
  The linear measurements of arch dimensions in millimeter before and after treatment with both methods of lip taping in both experimental groups
  Linear measurements for maxillary arch assessments in millimeters:
  * Antero-posterior arch length (I-ITT')
  * Posterior arch width (T-T')
  * Alveolar cleft widths (AP); Right cleft and (A'P') Left cleft
  * Mid-palatal arch width (C-C')
Assessment of Angular measurement change | T1 before starting any treatment and T2 After treatment before surgical repair (average 3 months)]
  The angular measurements of arch dimensions in degrees before and after treatment with both methods of lip taping in both experimental groups.
  Angular measurements for maxillary arch assessments in degrees:
  Anterior arch curvature angle (AIA')
Assessment of Parents Perception and experience | T1 before starting any treatment and T2 After treatment before surgical repair (average 3 months)]
  The perception and experience of parents of children with cleft lip and palate concerning the use presurgical infant orthopedics using a questionnaire-based cross-sectional survey. The assessment of mothers' perception and experience regarding PSIO will be executed using 15 validated preformed questions.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, Baghdad, Al-Rusaffa, Iraq

IPD SHARING:
Plan to Share IPD: No